CLINICAL TRIAL: NCT00309517
Title: A Prospectively Randomized Study on Neoadjuvant Radio-Chemotherapy in Patients With Operated Rectal Carcinoma Dukes B and C (pT2, pN1-3; pT3-4, pN0-3; M0.
Brief Title: Randomized Study on Neoadjuvant Radio-Chemotherapy in Rectal Carcinoma Dukes B and C
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABSCG 92
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2000-10

CONDITIONS: Rectal Cancer Dukes B, Dukes C
Keywords: Fluorouracil; Leucovorin; MAb 17-1A; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Leucovorin; Edrecolomab

INTERVENTIONS:
Drug: Fluourouracil
Drug: Leucovorin
Drug: MAb 17-1A

SUMMARY:
This clinical investigation examined the influence of preoperative radiotherapy in combination with postoperative 5-fluorouracil + leucovorin chemotherapy vs. 5-fluorouracil + leucovorin + MAb 17-1A chemo-immunotherapy on patients' local recurrence rate and overall survival time following surgery for rectal carcinoma Dukes B or C (T2-4, N0-3, M0).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically verified operable rectal cancer Dukes B and C (Stage II, T2-4, N0-3, M0), R0
* Age: 18-80 years
* Karnofsky Performance Status > 80
* Adequate bone marrow reserve (leukocytes > 4,000, thrombocytes > 105/mm3, Hb > 10g %), renal and hepatic functions (total bilirubin and creatinine < 1.25 x ULN)

Exclusion Criteria:

* Colon cancer
* R1, R2; carcinosis peritonei
* Start of treatment > 42 days postop; other adjuvant radiotherapy, chemotherapy or immunotherapy
* Previous application of a murine or chimeric monoclonal antibody or antibody fragment
* Medical therapy with steroids, cyclosporin or antithymocyte globulin within 3 months pre-study
* Known hypersensitivity to animal protein
* Serious concomitant disease: HIV, chronically inflammatory intestine, diabetes mell. gravis, cerebral seizure disorder, et al.
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 1997-07

PRIMARY OUTCOMES:
Local recurrence-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Jakesz, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group
Locations (8):
- Austria (8):
  - Hospital Oberpullendorf, Oberpullendorf, Burgenland
  - Hospital Baden, Baden, Lower Austria
  - Hospital Hainburg, Hainburg an der Donau, Lower Austria
  - Hospital Wiener Neustadt, Surgery, Wiener Neustadt, Lower Austria
  - Medical University of Graz, Oncology, Graz, Styria
  - General Hospital Linz, Linz, Upper Austria
  - Hospital BHB Linz, Linz, Upper Austria
  - Medical University of Vienna, General Hospital, Vienna, Vienna

REFERENCES:
- See also: Related Info — http://www.abcsg.at